CLINICAL TRIAL: NCT00147836
Title: Evaluation of the Effects of Oral Anti-Hyperglycemic Agents, Multiple Daily Injections or Continuous Subcutaneous Insulin Infusion on Glycemic Control, B-Cell Function and the Remission Rate in Newly-Diagnosed Type 2 Diabetic Patients
Brief Title: Evaluation of the Effects of Different Interventions on Glycemic Control in Newly-Diagnosed Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Education, China (Other Government); Guangdong Science and Technology Bureau, China (Unknown); Hoffmann-La Roche (Industry); Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NECT-2004-WJP; GSTB-05100981-LYB
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; therapy; sulfonylureas; metformin; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; Insulin, Isophane; Gliclazide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CSII (Active Comparator): Patients in continuous subcutaneous insulin infusion group received Human Insulin (Novolin-R, Novo Nordisk) with an insulin pump (H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland);
  Interventions: Drug: Human Insulin (Novolin-R, Novo Nordisk); Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland
- MDI (Active Comparator): Patients in MDI group were treated with pre-meal Novolin-R, and Human Insulin NPH (Novolin-N, Novo Nordisk) at bedtime. Initial insulin doses were 0.4-0.5 IU/kg and total daily doses were divided into 50% of basal and 50% of bolus injection in CSII group and 30%-20%-20%-30% in multiple daily insulin injection group
  Interventions: Other: Pre-meal; Drug: Novolin-R; Drug: Human Insulin NPH (Novolin-N, Novo Nordisk)
- OHA (Active Comparator): In oral hpoglycemic agents group, the patients with 20 kg/m2<BMI≤25kg/m2 were initiated with Gliclazide (Diamicron, Servier) 80mg Bid (maximum to 160mg Bid), the patients with 25kg/m2<BMI≤35kg/m2 were initiated with Metformin (Glucophage, BMS) 0.5 Bid (maximum to 2.0g/d), the combination of Diamicron and Glucophage was used in patients who could not achieve glycaemic control goal with one OHA or with FPG≥11.1mmol/l at randomization
  Interventions: Drug: Gliclazide (Diamicron, Servier); Drug: Diamicron and Glucophage

INTERVENTIONS:
Drug: Human Insulin (Novolin-R, Novo Nordisk)
  Arms: CSII
Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland
  Arms: CSII
Other: Pre-meal
  Arms: MDI
Drug: Novolin-R
  Arms: MDI
Drug: Human Insulin NPH (Novolin-N, Novo Nordisk)
  Arms: MDI
Drug: Gliclazide (Diamicron, Servier)
  Arms: OHA
Drug: Diamicron and Glucophage
  Arms: OHA

SUMMARY:
The purpose of this study is to investigate and evaluate the effects of different interventions (1.continuous subcutaneous insulin infusion,2.multiple daily injections, 3.anti-hyperglycemic agents) on glycemic control, B-cell function and the remission rate in newly-diagnosed type 2 diabetic patients.

DETAILED DESCRIPTION:
ß-Cell dysfunction and decreased insulin sensitivity are the main pathophysiological defects responsible for the development of hyperglycemia. With continuous presence of insulin resistance, progressive loss of ß-cell function is the crucial defect. Hyperglycemia has deleterious effect on β-cell function, which is partially reversible by adequate glycemic control. In newly diagnosed type 2 diabetic patients with severe hyperglycemia, 2 weeks continuous subcutaneous insulin infusion (CSII) can induce adequate glycemic control with improvement of β-cell function. Nearly half of the patients can maintain euglycemia longer than 12 months by transient CSII. The improvement of β-cell function, especially the restoration of the first-phase insulin response is related to sustained euglycemia in the newly diagnosed type 2 diabetic patients. But it is unclear whether any other interventions (such as oral hypoglycemic agents and multiple daily injections) inducing optimal glycemic control in a short period of time can have the same effect. As a multicenter, open-label, randomized, parallel-group study will be needed to further prove and clarify the findings.

ELIGIBILITY:
Inclusion Criteria:

1. informed consents be given before treatment
2. the newly-diagnosed type 2 diabetic patients
3. fasting blood glucose (FBG) level ranging from 7.0～16.7 mmol/L
4. age ranging from 25～70 years old
5. body mass index (BMI) ranging from20～35kg/m2
6. never be treated with any anti-hyperglycemic agents or anti-hyperlipidemic agents

Exclusion Criteria:

1. having any severe acute or chronic complications
2. renal dysfunction, blood creatinine≥150µmol/L
3. blood aminotransferase level rising up(more than 2 times of the normal level)
4. any severe cardiac disease including congestive cardiac failure, unstable angina and myocardial infarct in 12 months
5. serious hypertension (systolic pressure≥180mmHg and/ or diastolic pressure≥110mmHg)
6. chronic or acute pancreatic disease
7. severe systematic diseases or malignant tumor
8. allergic to the drugs using in the trial
9. any factors interfering the result
10. female patients incline to be pregnant
11. being treated with corticosteroid, immunosuppressing drugs or cytotoxic drugs
12. poor compliance

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
glycemic control, the improvement of β-cell l function and the remission rate after short intensive therapy in newly diagnosed type 2 diabetic patients | Oct. 2007

SECONDARY OUTCOMES:
the effects of different interventions (oral anti-hyperglycemic agents, multiple daily injections and continuous subcutaneous insulin infusion) on glycemic control, β-cell function and the remission rate in newly-diagnosed type 2 diabetic patients | Oct. 2007

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Weng, MD,PHD, Principal Investigator — Ministry of Education
Locations (1):
- the first Affiliated Hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Li Y, Xu W, Liao Z, Yao B, Chen X, Huang Z, Hu G, Weng J. Induction of long-term glycemic control in newly diagnosed type 2 diabetic patients is associated with improvement of beta-cell function. Diabetes Care. 2004 Nov;27(11):2597-602. doi: 10.2337/diacare.27.11.2597. PMID 15504992
- [Derived] Weng J, Li Y, Xu W, Shi L, Zhang Q, Zhu D, Hu Y, Zhou Z, Yan X, Tian H, Ran X, Luo Z, Xian J, Yan L, Li F, Zeng L, Chen Y, Yang L, Yan S, Liu J, Li M, Fu Z, Cheng H. Effect of intensive insulin therapy on beta-cell function and glycaemic control in patients with newly diagnosed type 2 diabetes: a multicentre randomised parallel-group trial. Lancet. 2008 May 24;371(9626):1753-60. doi: 10.1016/S0140-6736(08)60762-X. PMID 18502299